CLINICAL TRIAL: NCT04266769
Title: Precision Orthodontics: A Comparison of Custom vs Traditional Bracket Treatment Efficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LightForce Orthodontics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00040384
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Dental Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients with Malocclusion (Experimental)
  Interventions: Device: LightForce Orthodontic System

INTERVENTIONS:
Device: LightForce Orthodontic System — The LightForce Orthodontic System is a a digital treatment planning platform and patient-specific 3D printed polycrystalline alumina brackets for the treatment of malocclusion

SUMMARY:
This investigational testing aims to target multiple investigations sites to examine treatment efficiency metrics using a completely digital and patient-specific bracket treatment system for the correction of malocclusions.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be healthy and between the ages of 10 and 65.
* Eruption of all permanent teeth excluding second and third molars
* Sufficient labial tooth surface for bonding
* No more than one tooth missing from a single arch quadrant
* No existing molar tubes or bands

Exclusion Criteria:

* Presence of systemic diseases, cleft lip and palate, craniofacial anomalies, syndromes affecting bone or teeth, impacted teeth (excluding 3rd molars), and tumors of the parathyroid gland
* Presence of bridges or implants
* Cases requiring orthognathic surgery
* Significant periodontal disease
* Intake of drugs affecting tooth movement or bone formation (chronic use of Non-Steroidal Anti-Inflammatory Drugs, bisphosphonates, levothyroxine, or teriparatide drug class)
* Pregnancy

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Fafara, BS, Study Director — LightForce Orthodontics
Locations (1):
- Walt Orthodontics, Maple, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Malocclusion
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline metrics were not taken for the study population.
Arm/Group | Patients With Malocclusion
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 14
Time to Bond [Mean (Standard Deviation); unit: Minutes] — Data was not collected for patients at a baseline Population: Data was not collected for patients at a baseline
Length of treatment [Mean (Standard Deviation); unit: months] — Data was not collected for patients at a baseline Population: Data was not collected for patients at a baseline
length of debonding appointment [Mean (Standard Deviation); unit: Minutes] — Data was not collected for patients at a baseline Population: Data was not collected for patients at a baseline
length of time to achieve level and align [Mean (Standard Deviation); unit: months] — Data was not collected for patients at a baseline Population: Data was not collected for patients at a baseline
number of unscheduled appointments [Mean (Standard Deviation); unit: number of brackets] — Population: Data was not collected for patients at a baseline
Number of repositioned brackets [Mean (Standard Deviation); unit: number of brackets] — Population: Data was not collected for patients at a baseline

OUTCOME MEASURES:

1. Primary Outcome: Length of Bonding Appointment
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Patients With Malocclusion
Number analyzed (Participants) | 14
minutes | 33 (11)

2. Primary Outcome: Number of Debonded Brackets
Time Frame: approximately 2 years
Population: One patient did not complete treatment as they moved out of town and no longer went to the study's orthodontists.
Measure: Mean (Standard Deviation); unit: number of brackets
Arm/Group | Patients With Malocclusion
Number analyzed (Participants) | 13
number of brackets | 3 (2)

3. Primary Outcome: Length of Treatment
Time Frame: approximately 2 years
Population: One patient did not complete treatment as they moved out of town and no longer went to the study's orthodontists.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Patients With Malocclusion
Number analyzed (Participants) | 13
months | 27 (9)

4. Primary Outcome: Length of Debond Appointment
Time Frame: 1 day
Population: One patient did not complete treatment as they moved out of town and no longer went to the study's orthodontists.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Patients With Malocclusion
Number analyzed (Participants) | 13
minutes | 60 (0)

5. Primary Outcome: Length of Time to Achieve Leveling and Aligning
Time Frame: 2 years
Population: One patient did not complete treatment as they moved out of town and no longer went to the study's orthodontists.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Patients With Malocclusion
Number analyzed (Participants) | 13
months | 16 (7)

6. Primary Outcome: Number of Unscheduled Appointments
Time Frame: 2 years
Population: One patient did not complete treatment as they moved out of town and no longer went to the study's orthodontists.
Measure: Mean (Standard Deviation); unit: number of appointments
Arm/Group | Patients With Malocclusion
Number analyzed (Participants) | 13
number of appointments | 3 (2)

7. Primary Outcome: Number of Repositioned Brackets
Time Frame: 2 years
Population: One patient did not complete treatment as they moved out of town and no longer went to the study's orthodontists.
Measure: Mean (Standard Deviation); unit: number of brackets
Arm/Group | Patients With Malocclusion
Number analyzed (Participants) | 13
number of brackets | 1 (2)

ADVERSE EVENTS:
Time Frame: Patients were evaluated for any adverse events over their treatment, an expected average of 2 years. However, two patients had treatment times over 2 years with the maximum being under 4 years/
Arm/Group | Patients With Malocclusion
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT04266769/Prot_SAP_000.pdf